CLINICAL TRIAL: NCT01285245
Title: Effect of Interleukin-1 Receptor Antagonist on Insulin Sensitivity in Type 1 Diabetes Mellitus.
Brief Title: Effect of Anakinra on Insulin Sensitivity in Type 1 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Edwin J.P. van Asseldonk, Radboud University Nijmegen Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL34377.091.10; 2010-023479-24 (EudraCT Number)
Record Dates: First submitted 2010-11-26; First posted 2011-01-27 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes Mellitus
Keywords: insulin sensitivity; interleukin-1 receptor antagonist; inflammation; hyperglycemia-induced insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kineret (Experimental)
  Interventions: Drug: kineret

INTERVENTIONS:
Drug: kineret — once daily 100 mg of kineret subcutaneously for 8 days
  Other Names: anakinra; interleukin-1 receptor antagonist

SUMMARY:
The purpose of this study is to test whether anakinra is able to reduce insulin resistance.

This will be tested in overweighted type I diabetes mellitus patients, which have no residual beta-cell function. By using this patient group, all positive effects on glycemic control should be the consequence of improved insulin sensitivity.

DETAILED DESCRIPTION:
Although typically associated with type 2 diabetes, insulin resistance has been documented in Type 1 diabetes. Insulin resistance may also play an important role in the pathophysiology of type 1 diabetes mellitus. Once diabetes has emerged chronically elevated glucose levels further induce insulin resistance (glucose toxicity).

Inflammation is an important link between obesity and insulin resistance. The mechanism of hyperglycemia-induced insulin resistance is not clear, but evidently must be related to high glucose levels. There are indications that chronic hyperglycemia can induce inflammation, for example hyperglycemia induces IL-1β release, and recent studies have shown an interaction with thioredoxin interacting protein (TXNIP), at the level of the beta-cell but also, as found by our own group, at the level of the adipose tissue

All together, these findings suggest that blocking IL-1β-receptor activation by the interleukin-1 receptor antagonist anakinra, may reverse insulin resistance associated both with obesity and/or chronic hyperglycemia. When applied in (hyperglycemic) subjects with type 2 diabetes, blocking IL-1β should diminish the effects of glucose toxicity both at the level of beta-cell function as at the level of insulin sensitivity. When applied in (hyperglycemic) subjects with type 1 diabetes, the effects of glucose toxicity at the level of insulin sensitivity should decrease.

In order to be able to study an isolated effect of IL-1β blockade on insulin sensitivity, this study will test this hypothesis in subjects with type 1 diabetes and hence provide a proof of principle in vivo in humans for a proposed link between hyperglycemia, inflammation and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than 5 years
* Body mass index of > 25 kg/m2
* Insulin requirement > 0.5 U/kg bodyweight
* HbA1c>7.5%, stable glycemic control

Exclusion Criteria:

* Inability to give informed consent
* Presence of any medical condition that might interfere with the current study protocol.
* Immunodeficiency or immunosuppressive treatment (including TNFα blocking agents and corticosteroids)
* Anti-inflammatory drugs (including nonsteroidal anti-inflammatory drugs, 100 mg or less of aspirin per day is allowed)
* Signs of current infection (fever, C-reactive protein (CRP) > 30 mmol/l, treatment with antibiotics, previous or current diagnosis of tuberculosis.
* A history of recurrent infections
* Pregnancy or breast-feeding (contraception of at least 3 months before inclusion is required for fertile women)
* Liver disease (aspartate aminotransferase or alanine aminotransferase level of more than three times the upper limit of normal range)
* Renal disease (creatinine > 130 µmol/l
* Neutropenia < 2 x 109/l

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
insulin sensitivity as determined by euglycemic hyperinsulinemic clamp | change in insulin sensitivity after 1 week of treatment with anakinra as compared to baseline
  insulin sensitivity measured by euglycemic hyperinsulinemic clamp

SECONDARY OUTCOMES:
glycemic control | baseline, after 1 week of treatment and 4 weeks after treatment termination
  HbA1c, fasting glucose
adipocyte insulin sensitivity | baseline, after 1 week of treatment, 4 weeks after treatment termination
circulating hormonal and inflammatory factors and lipid profile | baseline, after 1 week of treatment, 4 weeks after treatment termination
insulin sensitivity as determined by euglycemic hyperinsulinemic clamp | change in insulin sensitivity 4 weeks after stopping anakinra treatment as compared to baseline
  insulin sensitivity measured by euglycemic hyperinsulinemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Cees J Tack, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands